CLINICAL TRIAL: NCT06818539
Title: Burnout in Hospital-based Nursing and Medical Personnel and Trainees: A Mixed Methods Approach
Brief Title: Burnout and Resilience in Hospital-based Nursing and Medical Personnel and Trainees
Acronym: RESIST
Status: Not yet recruiting | Type: Observational
Sponsor: University of Limerick (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Rigshospitalet, Denmark (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: EHSREC2024_06_02; KEEPCARING #101137244 (Other: EU)
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Stress; Burnout
Keywords: stress; burnout; resilience; crosssectional; healthcare workers; nurses; doctors; surgeons; observational; healthcare professionals; work stress
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Doctors and nurses: Hospital-based doctors and nurses, surgical as well as non-surgical pathways

SUMMARY:
Aims to look at associations between work stress, burnout and resilience in hospital-based nurses and medical professionals in several EU countries.

DETAILED DESCRIPTION:
Healthcare professionals, in particular, hospital-based nursing and medical staff, especially surgical specialities, are experiencing symptoms of burnout as never before. Within healthcare, job commitment is at stake leading to staff shortages which places further stress on the health care system, creating a vicious cycle of stressful work environment.

This is the context of the present study, and our aim is to explore quantitatively how factors like resilience, work-setting factors like job support, autonomy and leadership contribute to burnout in hospital-based nursing and medical personnel. These factors have been found to be predictive of burnout with few studies looking at synergistic interactions between these predictors. A survey design will be used for quantitative data collection. This study will also include qualitative interview-based study to complement the quantitative study.

ELIGIBILITY:
Inclusion Criteria:

* Hospital-based nurses and doctors

Exclusion Criteria:

* Non-hospital based healthcare professionals, under 18 and over 66, non-medical hospital staff

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital-based doctors and nurses across the European Union
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Resilience scores among hospital-based doctors and nurses | 5 months
  Resilience will be measured with Short Resilience Survey (SRS), an 8-item short resilience scale developed for healthcare workers. This measure consists of two subscales, Activation and Decompression. An examples of Decompression items include "can enjoy my personal time without focusing on work matters" and Activation "I care for all patients/clients equally even when it is difficult." These measures exist independent of employee engagement, indicating an empirical distinction between the two concepts. Response categories on the items (with 1 =Strongly Disagree to 5 = Strongly Agree), with higher scores indicating better Activation and Decompression ability.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gallagher, PhD, Principal Investigator — University of Limerick
Locations (1):
- Department of Psychology, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No
This is an anonymised data without participant identifiers, and investigating aggregate data and not individual participant data.

REFERENCES:
- [Background] Greville-Harris M, Withers C, Wezyk A, Thomas K, Bolderston H, Kane A, McDougall S, Turner KJ. Association of resilience and psychological flexibility with surgeons' mental wellbeing. BJS Open. 2024 Jul 2;8(4):zrae060. doi: 10.1093/bjsopen/zrae060. PMID 39041733
- [Background] Cha YJ, Lee KS, Cho JH, Choi IS, Lee D. Effect of Job Stress on Burnout among Nurses Responding to COVID-19: The Mediating Effect of Resilience. Int J Environ Res Public Health. 2022 Apr 29;19(9):5409. doi: 10.3390/ijerph19095409. PMID 35564803
- [Background] Morgan KH, Libby NE, Weaver AK, Cai C. Development of an early warning resilience survey for healthcare organizations. Heliyon. 2019 Nov 1;5(10):e02670. doi: 10.1016/j.heliyon.2019.e02670. eCollection 2019 Oct. PMID 31720458
- See also: This study is part of a larger EU-funded project called KEEPCARING: Future Proofing Health- and Care Systems Safeguarding Healthcare Workers in Hospital Settings. — https://keepcaring.eu/

DOCUMENTS (2):
  • Study Protocol (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT06818539/Prot_000.pdf
  • Informed Consent Form (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/39/NCT06818539/ICF_001.pdf